CLINICAL TRIAL: NCT02700854
Title: Hypoxic-Ischemic Encephalopathy Therapy Optimization for Better Neuroprotection With Inhalative CO2 in Asphyxiated, Cooled, Mechanically Ventilated Neonates at Risk for Hypocapnia
Brief Title: Hypoxic-Ischemic Encephalopathy Therapy Optimization in Neonates for Better Neuroprotection With Inhalative CO2
Acronym: HENRIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Ágnes Jermendy, assistant lecturer, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1Ped-AsphHENRIC001
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Hypoxic-Ischaemic Encephalopathy; Perinatal Asphyxia; Hypocapnia
Keywords: Hypothermia treatment; Hypocapnia; Inhaled CO2; Neuroprotection
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypocapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5% carbon-dioxide inhalation (Experimental): 5% carbon-dioxide will be administered through patient circuits to asphyxiated, cooled, mechanically ventilated newborns at risk for hypocapnia
  Interventions: Other: 5% carbon-dioxide inhalation

INTERVENTIONS:
Other: 5% carbon-dioxide inhalation — 5% CO2 (36 mmHg) and 95% air gas mixture inhalation, for a maximum of 12 hours or until metabolic acidosis recovery occurs as measured by BE > -5 mmol/L in arterial blood gas samples
  Other Names: N-Carbogen

SUMMARY:
This is a Phase I, open-label, single center trial to evaluate the feasibility and safety of low concentration CO2 gas mixture (5% CO2 + 95% air) inhalation in asphyxiated, cooled, mechanically ventilated newborns at risk of hypocapnia with The hypothesis is that hypocapnia, which is driven by hyperventilation in the presence of metabolic acidosis, is deleterious to the injured brain and can be safely avoided with low concentration CO2 inhalation.

DETAILED DESCRIPTION:
Specific aims:

1. To test the feasibility of low concentration inhalative CO2 gas mixture (5% CO2 + 95% air) administration to achieve a desired range of pCO2 of 40-60 mmHg in asphyxiated, cooled, mechanically ventilated newborns at risk of hypocapnia with moderate to severe hypoxic-ischemic encephalopathy.
2. To test the safety of CO2 gas mixture (5% CO2 + 95% air) inhalation in asphyxiated, cooled, mechanically ventilated newborns at risk of hypocapnia with moderate to severe hypoxic-ischemic encephalopathy.

Term infants (≥ 36 weeks of gestation) will have to be at risk of hypocapnia to be eligible, as defined by a temperature corrected pCO2 ≤ 40 mmHg in blood gas analysis, at any time within six hours of life.

The gas mixture will be administered through patient circuits in conventional ventilators. Administered CO2 level will be closely monitored at the inhalation circuit (constant 5% = 36 mmHg). Blood gas samples will be taken hourly to ensure targeted and tolerable pCO2 levels.

ELIGIBILITY:
Inclusion Criteria:

* At any time within six hours of life the temperature corrected pCO2 is less than or equal to 40 mmHg after the parameters of mechanical ventilation is set according to standard protocol (SIMV+VG 5ml/kg, fr 20/min, PEEP 5 H20cm, Ti 0,35-0,45 sec).
* Moderate hypoxic- ischaemic encephalopathy, fulfilling TOBY criteria (A, B, C).
* ≥ 36. gest. week
* < 6th hours of life
* Hypothermia treatment
* Parental consent form
* Spontaneous breathing
* Endotracheal intubation
* AUC, VUC in place

Exclusion Criteria:

* Major birth defect
* Meconium aspiration syndrome
* Need for combined catecholamine therapy
* FiO2 > 40%
* Htc < 35%
* Acid-base status: pH < 6.8, lactate > 15mM
* Excessive bicarbonate administration during initial stabilization (> 1mmol/kg)

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the desired pCO2 range of 40-60 mmHg (temp. corrected) during CO2 inhalation. | 3 days

SECONDARY OUTCOMES:
Number of seizures, either detected clinically or by amplitude integrated EEG monitoring | Within one week
Time until the end point of metabolic acidosis (BE > -5 mmol/L) | During CO2 inhalation (max. 12 hours)
Time until the end point of acidosis (pH > 7.25) | During therapeutic hypothermia (max. 72 hours)
Severe hypotension (mean arterial pressure less than 25 mmHg), despite full inotrope support and volume replacement. | During therapeutic hypothermia (max. 72 hours)
Intracranial haemorrhage detected by MRI | Within seven days
Reduction in Lac/NAA ratio on magnetic resonance spectroscopy | Within seven days
Preserved fractional anisotropy measured on diffusion weighted MRI | Within seven days
Death | Within one month

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Szabó, MD, PhD, Study Director — Semmelweis University, 1st Department of Pediatrics
Locations (1):
- Semmelweis University, 1st Department of Pediatrics, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laffey JG, Kavanagh BP. Hypocapnia. N Engl J Med. 2002 Jul 4;347(1):43-53. doi: 10.1056/NEJMra012457. No abstract available. PMID 12097540
- [Background] Pappas A, Shankaran S, Laptook AR, Langer JC, Bara R, Ehrenkranz RA, Goldberg RN, Das A, Higgins RD, Tyson JE, Walsh MC; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Hypocarbia and adverse outcome in neonatal hypoxic-ischemic encephalopathy. J Pediatr. 2011 May;158(5):752-758.e1. doi: 10.1016/j.jpeds.2010.10.019. Epub 2010 Dec 10. PMID 21146184
- [Background] Klinger G, Beyene J, Shah P, Perlman M. Do hyperoxaemia and hypocapnia add to the risk of brain injury after intrapartum asphyxia? Arch Dis Child Fetal Neonatal Ed. 2005 Jan;90(1):F49-52. doi: 10.1136/adc.2003.048785. PMID 15613575
- [Background] Azzopardi DV, Strohm B, Edwards AD, Dyet L, Halliday HL, Juszczak E, Kapellou O, Levene M, Marlow N, Porter E, Thoresen M, Whitelaw A, Brocklehurst P; TOBY Study Group. Moderate hypothermia to treat perinatal asphyxial encephalopathy. N Engl J Med. 2009 Oct 1;361(14):1349-58. doi: 10.1056/NEJMoa0900854. PMID 19797281